CLINICAL TRIAL: NCT02951871
Title: Causes of Death in Follicular Lymphoma: a Single Center Retrospective Analysis
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0719
Record Dates: First submitted 2016-10-31; First posted 2016-11-01 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-10

CONDITIONS: This Study Describes the Different Causes of Death in 237 FL Patients
Keywords: Follicular lymphoma; death, rituximab, treatment related toxicity
MeSH Terms: conditions — Lymphoma, Follicular; Death

STUDY DESIGN:
Time Perspective: Retrospective

GROUPS / COHORTS (4):
- LP: Lymphoma Progression
- TRM: Treatment Related Mortality
- NHM: Non hematologic malignancy
- OC: Other Cause

SUMMARY:
Background.Although the life expectancy of patients with FL has recently increased, notably since the introduction of rituximab in combination with chemotherapy, little is known regarding the precise causes of patients death. Patients and methods'. This study describes the different causes of death in FL patients among followed since 2000 at Lyon University Hospital, centre Léon Bérard and Mayo Clinic. The causes of death will be classified as related to lymphoma progression, treatment-related toxicity (including TRM and secondary myelodysplastic syndrome/acute myeloid leukemia), secondary neoplasias, or other.

ELIGIBILITY:
Inclusion Criteria:

* FL patients
* patients recorded as deceased

Exclusion Criteria:

-Other diagnosis than FL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective analysis was performed in 3 reference center where patients were treated and regularly followed for FL between January 2000 and December 2015. All patients were initially staged according to the conventional recommendations, including a clinical examination and blood tests, a bone marrow biopsy, and a computerized tomography body scan. The treatment modalities have evolved over time and were chosen according to the institutional guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2000-01; Primary Completion 2016-01 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
overall survival (OS) | OS length was calculated from the date of diagnosis to the date of death

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier Lyon sud, Pierre-Bénite, Auvergne-Rhône-Alpes, France